CLINICAL TRIAL: NCT05910502
Title: Autism Family Empowerment Coaching and Training Program (AFECT): Evaluating a Parent Coaching and Family Navigation Program for New Autism Spectrum Disorder Diagnosis
Brief Title: Project AFECT (Autism Family Empowerment Coaching and Training Program)
Acronym: AFECT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Heidi M. Feldman, Professor of Developmental and Behavioral Pediatrics, Stanford University School of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB#69103
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder; Autism; Autism Spectrum Disorders; Autistic Disorder; Autistic Spectrum Disorder; Autistic Spectrum Disorders; Autistic Disorders Spectrum
Keywords: Parent Coaching; Family Navigation; Parent Training; Parent Stress; Parent Self-Efficacy; Service Navigation
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Child Development Disorders, Pervasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coaching Group (Experimental): Coaching Group will receive Project AFECT intervention, in addition to treatment as usual.
  Interventions: Behavioral: Autism Family Empowerment Coaching and Training Program

INTERVENTIONS:
Behavioral: Autism Family Empowerment Coaching and Training Program — Participants in the intervention group will be connected with Project AFECT Coaches who will provide: Coaching to (1) assure parents understand diagnosis, (2) assist parents in finding accurate, current information about autism, (3) guide parents to free online autism training resources, (4) empower parents to evaluate child's intervention plan holistically, and (5) provide emotional support to reduce stress; Navigation to (1) help family access autism treatments, and (2) connect to early intervention and educational services.
  Other Names: Project AFECT

SUMMARY:
The goal of this clinical trial is to learn about the journey of families after their child's diagnosis of autism and to help parents understand autism and get the right treatments for their child. This study is for parents of children just diagnosed with autism who are:

* Age greater than 1 and up to 5 years old;
* Hispanic/Latino OR Black/African-American OR have Medi-Cal as primary health insurance; AND
* Live in one of the following counties in California (Alameda, Contra Costa, Marin, Monterey, Napa, San Benito, San Francisco, San Mateo, Santa Clara, Santa Cruz, Solano, or Sonoma).

The main questions it aims to answer are:

* Whether parent coaching through Project AFECT leads to decreased parental stress and increased parental confidence;
* Whether family navigation through Project AFECT leads to increased number of referrals to early intervention and educational services and reduced wait times to autism treatments;
* Whether children whose parents receive Project AFECT intervention show increased language skills compared to children whose parents did not receive intervention.

Participants will be asked to:

* Complete surveys at enrollment and 3 and 6 months later.
* Work with Project AFECT Coach.

Researchers will compare control and intervention groups to see if Project AFECT leads to improved parent and child outcomes.

DETAILED DESCRIPTION:
This is a prospective clinical effectiveness study of Project AFECT, an intervention combining parent coaching and family navigation. Parents who meet inclusion criteria will be invited to participate in this study at the time of their child's autism diagnosis at Stanford Medicine Children's Health.

In addition to treatment as usual, participants in the intervention group will be connected with Project AFECT Coaches who will provide: Coaching to (1) assure parents understand diagnosis, (2) assist parents in finding accurate, current information about autism, (3) guide parents to free online autism training resources, (4) empower parents to evaluate child's intervention plan holistically, and (5) provide emotional support to reduce stress; Navigation to (1) help family access autism treatments, and (2) connect to early intervention and educational services.

ELIGIBILITY:
Inclusion Criteria:

1. Parents of children just diagnosed with autism (with or without other diagnoses) who are:

1. Age greater than 1 and up to 5 years old;
2. Hispanic/Latino OR Black/African-American OR have Medi-Cal as primary health insurance; AND
3. Live in one of the following counties in California (Alameda, Contra Costa, Marin, Monterey, Napa, San Benito, San Francisco, San Mateo, Santa Clara, Santa Cruz, Solano, or Sonoma).

Exclusion Criteria:

* Non-legal guardians or foster parents who provide care to children newly diagnosed with autism.
* Parents of children without diagnosis of autism.

Ages: 12 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-Efficacy | From enrollment to the end of intervention at 6 months
  Mean change from baseline in parental self-efficacy measured using Autism-Specific Parenting Self-Efficacy Scale (PSEaS). Overall possible scores on the scale range from 17 - 85. The higher the score, the higher the measured level of parental self-efficacy (better outcome).
Stress Level | From enrollment to the end of intervention at 6 months
  Mean change from baseline in parental stress level measured using Parental Stress Scale (PSS). Overall possible scores on the scale range from 18 - 90. The higher the score, the higher the measured level of parental stress (worse outcome).

SECONDARY OUTCOMES:
Child's Language Development | From enrollment to the end of intervention at 6 months
  Scores using MacArthur-Bates Communicative Development Inventory - Words and Gestures. For comparison between groups, we will be utilizing the raw scores. Overall possible raw scores range from 0 - 396. The higher the raw score, the higher the number of words understood and produced by the child (better outcome).
Access to autism treatments | From enrollment to the end of intervention at 6 months
  Time from initial autism diagnosis to start of applied behavior analysis (ABA) therapy
Access to early intervention/special education | From enrollment to the end of intervention at 6 months
  Time from initial autism diagnosis to assessment for early intervention/special education and development of Individualized Family Service Plan (IFSP)/Individualized Education Program (IEP)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Feldman, MD, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Gardner Packard Children's Health Center, Atherton, California
  - Stanford Medicine Children's Health, Sunnyvale, California

IPD SHARING:
Plan to Share IPD: Yes
After conclusion of this study and publication of the main findings, de-identified data will be placed in a public repository.